CLINICAL TRIAL: NCT02342977
Title: Effects of Lacosamide on Post-operative Opioid Requirements After a Total Hip Arthroplasty: A Randomized Double -Blinded, Placebo-controlled Pilot Study.
Brief Title: Effects of Lacosamide on Post-operative Opioid Requirements After a Total Hip Arthroplasty:
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: We were unable to enroll any patients into the study.
Sponsor: Indiana University School of Medicine (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bryan Sakamoto, Effects of lacosamide on post-operative opioid requirements after a total hip arthroplasty: A randomized double -blinded, placebo-controlled pilot study., VA Office of Research and Development
Organization: Indiana University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1408905316
Record Dates: First submitted 2014-12-18; First posted 2015-01-21 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Avascular Necrosis
Keywords: total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patient will randomly receive a placebo
  Interventions: Drug: Placebo
- Experimental (Experimental): Patients will randomly receive experimental drug (lacosamide).
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Placebo — Patients will randomly receive placebo
  Arms: Placebo
Drug: Lacosamide — Patients will randomly receive lacosamide
  Arms: Experimental

SUMMARY:
The purpose of this study is to determine how effect lacosamide is in reducing the amount of pain medication needed following a total hip arthroplasty. The study team hypothesizes that a single dose of lacosamide will reduce the amount of pain medication required after surgery. The study team plans to evaluate the amount of pain medication needed and quality of pain control during a subject's hospital stay and at their three month follow-up visit following their surgery.

DETAILED DESCRIPTION:
All patients who agree to participate in this study will receive the same surgical and anesthetic techniques that are provided to all our patients undergoing this procedure at this institution. Post-operative treatment and therapy and follow-up will also be the same as any of our patients undergoing this procedure at this institution.

The only difference would be that patients would be randomized (determined by chance, like a flip of a coin) to either receive a single dose of lacosamide (100 mg by mouth) or placebo (sugar pill by mouth) before the surgical procedure. This would be the only experimental part of this study.

In addition, specific information will be collected throughout the patients care until discharged from the orthopedic clinic (approximately 3 months after the procedure). The collected information will include subject's age, race and ethnicity, sex, height, weight, American Society of Anesthesiologist physical status, total amount of opioid (pain medication) use, pain scores, nausea and vomiting, time spent in the post anesthesia care unit (time to discharge readiness), and discharge from the hospital. The patient's pain score and opioid use will be assessed during their follow-up at approximately 3 months (Note: all of the specific information collected is normally gathered or documented in our surgical patients' record). In addition, participants may withdraw from the study at any time.

The main goal of this study is to determine if lacosamide can reduce the amount of opioids required in patient's undergoing a total hip arthroplasty. Lacosamide is a FDA approved medication for the treatment of partial-onset seizures and is a man-made amino acid (usually are used as the building blocks from which proteins are made in the body) which block special proteins inby a change in the electricity that a cell may feel (voltage-gated sodium channel). Lacosamide is a new antiepileptic drug apparently lacking any major pharmacokinetic interactions (how the body affects a specific drug after administration, as well as the chemical changes of the substance in the body, and the effects and routes of excretion of the metabolites of the drug).

Lacosamide, carbamazepine and oxcarbazepine are known to block special proteins in the covering of cells which allow sodium into the cells when they are turned on by a change in the electricity that a cell may feel (voltage-gated sodium channel, NaV1.7). Lacosamide was chosen over carbamazepine and oxcarbazepine because it causes fewer side effects. Currently, lacosamide is being tested in patients with painful diabetic nerve pain. Further trials to identify lacosamide's potential in pain control and for other indications have been started.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for participation if they are 18-70 years of age.
* Patients who have an American Society of Anesthesiologists physical status I-III.
* Patients who are scheduled for primary total hip arthroplasty.
* Any patients who are willing to comply with study requirements and agrees to be in the study.

Exclusion Criteria:

* A patient's refusal to participate.
* Inability to give consent.
* Any patients on a scheduled opioid regimen for pain greater than 3 months.
* Bleeding diathesis.
* Hypersensitivity to lacosamide or any component of the formulation (some formulation contains phenylalanine) and/or any drug allergies to any medications used in this study.
* Second- or third-degree atrioventricular (AV) block, sick sinus syndrome without pacemaker, sodium channelopathies (e.g., Brugada syndrome), myocardial ischemia, heart failure, and structural heart disease.
* Severe hepatic and or renal impairment.
* Pregnant or can become pregnant.
* Breast-Feeding.
* Have any suicidal thoughts, depression, or behavioral changes.
* Taking any antiepileptic medications.
* Any known seizure disorder (e.g. Lennox-Gastaut syndrome).
* Currently prescribed:

Carbamazepine Strong inhibitors of cytochrome P450-2C9 (Capecitabine; Delavirdine; floxuridine; Fluorouracil (Systemic); Gemfibrozil; Nicardipine; Sitaxentan; Sulfadiazine; Sulfissoxazole; Tegafur; Tolbutamide) Strong inhibitors of cytochrome P450-3A4 (Atazanavir; Boceprevir; Chloramphenicol; Clarithromycin; Cobicistat; Conivaptan; Darunavir; Delavirdine; Fosamprenavir; Indinavir; Itraconazole; Ketoconazole (Systemic); Lopinavir; Nefazodone; Nelfinavir; Nicardipine; Posaconazole; Ritonavir; Saquinavir; Telaprevir; Telithromycin; Voriconazole) Delavirdine Fosphenytoin Nicardipin Phenobarbital Phenytoin Ethinylestradiol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Opioid use in Post anesthesia care unit | 30 minutes to 2 hours after surgery
  Post operative opioid use.

SECONDARY OUTCOMES:
Pain scores | Post operative Day #0 through hospital discharge (4 day average)
  Post operative pain scores
Nausea and Vomiting | Post operative Day #0 through hospital discharge (4 day average)
  Post operative nausea and vomiting
Total opioid use | Post operative Day #0 through hospital discharge (4 day average)
  Total post operative opioid use
Time to PACU discharge readiness | 30 minutes to 2 hours after surgery
  Post operative discharge readiness
Pain scores and opioid use at 3 month discharge | At 3 month surgery follow up
  Development of chronic pain
Time to hospital discharge | Post operative Day #0 through hospital discharge ( 4 day average )
  Hospital discharge
Possible side effects from Lacosamide | Post operative Day #0 through hospital discharge (4 day average)
  Possible side effects ( dizziness, headaches, visual changes, and nausea )

CONTACTS AND LOCATIONS:
Overall Officials: Bryan M Sakamoto, M.D., PhD, Principal Investigator — Richard L. Roudebush VA Medical Center
Locations (1):
- Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana, United States